CLINICAL TRIAL: NCT00484133
Title: Microcirculation Guided Therapy Versus "Standard Treatment" of Severe Sepsis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: R. van Raalte, Onze Lieve Vrouwe gasthuis
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WO-06.068
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Last update posted 2008-01-22 (Estimated); Status verified 2008-01

CONDITIONS: Severe Sepsis; Microcirculation
Keywords: sepsis; severe sepsis; microcirculation; Orthogonal polarisation spectral
MeSH Terms: conditions — Sepsis | interventions — Dopamine; Dobutamine; Enoximone; Nitroglycerin; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dopamine
Drug: dobutamine
Drug: enoximone
Drug: nitroglycerine
Drug: noradrenaline

SUMMARY:
The purpose of this study is to asses the recovery of organ failure between two resuscitation protocols in severe sepsis: standard, pressure guided therapy versus a microcirculation guided therapy

DETAILED DESCRIPTION:
Despite continued improvements in medical therapy, mortality from septic shock has remained between 30% and 70% for the past three decades with only a slight decrease in mortality rate. Standard treatment of septic shock is fluid resuscitation, followed by agents with vasopressor activity to correct hypotension in septic shock. The question rises whether vasopressors should be the first line of action in septic shock Opening and recruiting the microcirculation are expected to improve regional organ function and tissue distress in severe sepsis. Beside fluid resuscitation, vasodilatation, in this respect, enhances microcirculatory flow while vasoconstriction causes a reduction in microcirculatory flow. On the other hand, a minimal perfusion pressure should be present. Our aim is to asses the effects of two resuscitation protocols in severe sepsis: the "standard treatment" using predefined pressure goals versus a microcirculation guided therapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* admission to the intensive care unit with severe sepsis, defined in according with a modification of the American College of Chest Physician/SCCM guidelines criteria
* intention to provide full intensive care treatment for at least 72 hours and
* written informed consent to be obtained from patient or next of kin.

Exclusion Criteria:

* haematologic malignancy
* metastatic malignancy
* AIDS with CD4 < 50 cells/mm3
* liver cirrhosis Child Pugh B & C
* pregnancy
* post resuscitation with GCS < 8 of 15 and treatment with induced hypothermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Difference in SOFA (Sequential Organ Failure Assessment) score during the first 72 hours of treatment for severe sepsis | 72 hours

SECONDARY OUTCOMES:
Severity, decrease and duration of organ failure over the complete ICU stay | complete icu stay
Duration of organ support | during ICU treatment
ICU and hospital length of stay | hospital stay
ICU and hospital mortality | hospital stay
Inflammatory response measured by IL-6/IL-10 | 72 hours
Plasma concentration of asymmetric dimethyl arginine (ADMA | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rutger v Raalte, MD, Principal Investigator — Onze Lieve Vrouwe Gasthuis, intensive care unit
Locations (1):
- Onze Lieve Vrouwe Gasthuis, intensive care, Amsterdam, Netherlands

REFERENCES:
- [Derived] van der Voort PH, van Zanten M, Bosman RJ, van Stijn I, Wester JP, van Raalte R, Oudemans-van Straaten HM, Zandstra DF. Testing a conceptual model on early opening of the microcirculation in severe sepsis and septic shock: a randomised controlled pilot study. Eur J Anaesthesiol. 2015 Mar;32(3):189-98. doi: 10.1097/EJA.0000000000000126. PMID 25032942